CLINICAL TRIAL: NCT03611309
Title: A Multi-Center Randomized Controlled Trial of Perioperative Palliative Care Surrounding Cancer Surgery for Patients and Their Family Members (the PERIOP-PC Trial)
Brief Title: Perioperative Palliative Care Surrounding Cancer Surgery for Patients & Their Family Members
Acronym: PERIOP-PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Karl Lorenz, Professor of Medicine (Primary Care and Population Health), Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-45805; NCI-2018-02183 (Other: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2018-07-25; First posted 2018-08-02 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Gastrointestinal Cancer
Keywords: Pancreatic Cancer; Hepatocellular Cancer; Esophageal Cancer; Gastric Cancer; Cholangio carcinomas
MeSH Terms: conditions — Gastrointestinal Neoplasms; Pancreatic Neoplasms; Liver Neoplasms; Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgeon-palliative care team co-management (Experimental): In the Surgeon-palliative care team co-management arm, all patients receive the surgical care of surgeon alone management, which includes surgeon and the surgical team. In addition to this surgeon alone care, palliative care will also be provided by a specialist team. For patients in this arm, patients and/or family members will be seen by the palliative care team: (1) in an outpatient setting prior to surgery, (2) in the hospital within 72 hours of their initial surgery and as needed afterwards, and (3) via phone on in-clinic (per patient preference) on an at least monthly basis and/or as needed for 12 weeks following surgery.
  Interventions: Other: Surgeon-palliative care team co management
- Surgeon alone management (Other): The surgeon and surgical team will manage symptoms, psychosocial support, and prognostic related communication. The surgeon and surgical team care for the patient and their family both prior to and following surgery. The surgeon team is given guidelines published by the National Cancer Coalition Network as to when palliative care specialist consultation is recommended
  Interventions: Other: Surgeon team alone management

INTERVENTIONS:
Other: Surgeon-palliative care team co management — Surgeon-palliative care team co management includes surgeon alone care and palliative care specialist team
  Arms: Surgeon-palliative care team co-management
Other: Surgeon team alone management — The surgeon and surgical team will manage
  Arms: Surgeon alone management

SUMMARY:
The study goal is to compare surgeon-palliative care team co-management, versus surgeon alone management, of patients and family members preparing for major upper gastrointestinal cancer surgery. The study also aims to explore, using qualitative methods, the impact of surgeon-palliative care team co-management versus surgeon alone management on the perioperative care experience for patients, family members, surgeons, and palliative care clinicians.

DETAILED DESCRIPTION:
The components of surgeon palliative care team co management practices will include Time, Education, Assessments, and Multi disciplinary (TEAM) element.

1. Time; At least 60 minutes/month (per patient and caregiver preference) devoted to palliative care treatments for the patient and family
2. Education - Patients and family members, per their desires and wishes, are counseled and educated about their disease, including self-management of symptoms, prognosis, and treatment options
3. Assessment - Formal assessment of symptoms including pain, dyspnea, constipation/diarrhea, anxiety/depression, fatigue, and nausea. Edmonton symptom score33 will be used as a formal assessment.
4. Multi-Disciplinary - Management must be multi disciplinary with access to a multi-disciplinary palliative care team composed of nurse, physician, social worker, pharmacist, and/or chaplain team members.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and must be able to give informed consent.
* Diagnosed with pancreatic cancer or hepatocellular cancer or esophageal cancer or gastric cancer and/or cholangio carcinomas
* Non emergent, upper gastrointestinal cancer related surgery with a goal of primary resection of the tumor- optimal surgical goal is cure, not merely disease palliation.
* One companion per patient will be allowed to participate. In addition, to being identified by the patient at being a key caregiver throughout the surgery period, these companions must be able to give informed consent and at least 18 years of age.

Exclusion Criteria:

* No previous involvement of palliative care providers in their care course

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl Lorenz, MD, MSHS, Principal Investigator — Stanford University
Locations (5):
- United States (5):
  - Stanford University, Stanford, California
  - Johns Hopkins Hostpital, Baltimore, Maryland
  - Dana Farber/ Brigham, Boston, Massachusetts
  - University of New Mexico, Albuquerque, New Mexico
  - Ohio State University Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holdsworth LM, Siden R, Lessios AS, Verano M, Rickerson E, Fahy B, Johnston FM, Waterman B, Aslakson R. Patient Experiences of Specialty Palliative Care in the Perioperative Period for Cancer Surgery. J Pain Symptom Manage. 2024 Sep;68(3):292-298.e1. doi: 10.1016/j.jpainsymman.2024.06.008. Epub 2024 Jun 19. PMID 38906425
- [Derived] Aslakson RA, Rickerson E, Fahy B, Waterman B, Siden R, Colborn K, Smith S, Verano M, Lira I, Hollahan C, Siddiqi A, Johnson K, Chandrashekaran S, Harris E, Nudotor R, Baker J, Heidari SN, Poultsides G, Conca-Cheng AM, Cook Chapman A, Lessios AS, Holdsworth LM, Gustin J, Ejaz A, Pawlik T, Miller J, Morris AM, Tulsky JA, Lorenz K, Temel JS, Smith TJ, Johnston F. Effect of Perioperative Palliative Care on Health-Related Quality of Life Among Patients Undergoing Surgery for Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2023 May 1;6(5):e2314660. doi: 10.1001/jamanetworkopen.2023.14660. PMID 37256623
- [Derived] Aslakson RA, Chandrashekaran SV, Rickerson E, Fahy BN, Johnston FM, Miller JA, Conca-Cheng A, Wang S, Morris AM, Lorenz K, Temel JS, Smith TJ. A Multicenter, Randomized Controlled Trial of Perioperative Palliative Care Surrounding Cancer Surgery for Patients and Their Family Members (PERIOP-PC). J Palliat Med. 2019 Sep;22(S1):44-57. doi: 10.1089/jpm.2019.0130. PMID 31486730

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 20 patients were discovered to have improperly filled out consents and could not be contacted to correct consent. The site's IRB determined that these patients be unenrolled from the study and that any data collected not be used.
Groups:
- Surgeon-palliative Care Team Co-management (Intervention): In the Surgeon-palliative care team co-management arm, all patients receive the surgical care of surgeon alone management, which includes surgeon and the surgical team. In addition to this surgeon alone care, palliative care will also be provided by a specialist team. For patients in this arm, patients and/or family members will be seen by the palliative care team: (1) in an outpatient setting prior to surgery, (2) in the hospital within 72 hours of their initial surgery and as needed afterwards, and (3) via phone on in-clinic (per patient preference) on an at least monthly basis and/or as needed for 12 weeks following surgery.
  Surgeon-palliative care team co management: Surgeon-palliative care team co management includes surgeon alone care and palliative care specialist team
- Surgeon Alone Management (Control): The surgeon and surgical team will manage symptoms, psychosocial support, and prognostic related communication. The surgeon and surgical team care for the patient and their family both prior to and following surgery. The surgeon team is given guidelines published by the National Cancer Coalition Network as to when palliative care specialist consultation is recommended
  Surgeon team alone management: The surgeon and surgical team will manage
Period: Overall Study
Arm/Group | Surgeon-palliative Care Team Co-management (Intervention) | Surgeon Alone Management (Control)
Started | 182 | 177
Completed | 161 | 162
Not Completed | 21 | 15
Not completed — Lost to Follow-up | 16 | 8
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Surgeon-palliative Care Team Co-management (Intervention) | Surgeon Alone Management (Control) | Total
Number analyzed (Participants) | 182 | 177 | 359
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Participants that reported their age are included in the analysis
  years
    number analyzed (Participants) | 181 | 176 | 357
    (all) | 64.57 (10.90) | 64.72 (10.40) | 64.66 (54.02)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 109 | 85 | 194
  Female | 73 | 90 | 163
  Unknown | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 18 | 41
  Not Hispanic or Latino | 159 | 157 | 316
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 2 | 7
  Asian | 4 | 9 | 13
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 11 | 16 | 27
  White | 145 | 136 | 281
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 14 | 13 | 27
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 182 | 177 | 359

OUTCOME MEASURES:

1. Primary Outcome: Patient Quality of Life Patient Quality of Life 12 Weeks After Surgery
Description: Patient quality of life will be measured by the Functional Assessment of Chronic Illness Therapy Palliative care subscale (FACIT-PAL). FACIT-PAL is a compilation of general questions divided into four primary QOL domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, and Functional Well-Being. FACIT-PAL has 46 item self report measure. The range is from 0-184 for the FACIT-PAL. A higher score is a better outcome.
Time Frame: Up to 12 weeks after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Surgeon-palliative Care Team Co-management | Surgeon Alone Management
Number analyzed (Participants) | 152 | 147
score on a scale | 138.54 (28.28) | 136.90 (28.96)
Statistical Analysis 1: Comparison: Surgeon-palliative Care Team Co-management vs Surgeon Alone Management; Test type: Superiority; p = .623, Regression, Linear — The a priori threshold for statistical significance was < 0.05; Mean Difference (Final Values) = -1.63, 95% CI 2-sided [-8.15 to 4.89] — FACIT-Pal Total score

2. Secondary Outcome: Patient Mood Symptoms Assessment 12 Weeks After Surgery
Description: Patient symptoms were measured using the Patient-Reported Outcomes Measurement Information System (PROMIS-29) version 2.1. PROMIS-29 survey questions were each rated on a 5-point Likert scale (range: 1 to 5, higher scores represent a better outcome). Item responses were converted to PROMIS T-scores per the PROMIS scoring manual (population mean = 50, SD = 10). T-scores were then converted to standardized z-scores using the formula (T-score - 50) / 10. Composite physical and mental health z-scores were calculated using weighted domain z-scores. Higher z-scores indicate better outcomes, and negative z-scores indicate scores below the population reference mean.
Time Frame: Up to 12 weeks after surgery
Population: Participants with available survey data
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Surgeon-palliative Care Team Co-management | Surgeon Alone Management
Number analyzed (Participants) | 144 | 145
z-score
  Physical health | -0.50 (1.01) | -0.43 (0.89)
  Mental health | -0.07 (0.84) | -0.07 (0.87)
Statistical Analysis 1: Comparison: Surgeon-palliative Care Team Co-management vs Surgeon Alone Management; Analysis of physical health score; Test type: Superiority; p = .555, Regression, Linear — The a priori threshold for statistical significance was < 0.05; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.29 to 0.15]
Statistical Analysis 2: Comparison: Surgeon-palliative Care Team Co-management vs Surgeon Alone Management; Analysis of mental health score; Test type: Superiority; p = .983, Regression, Linear — The a priori threshold for statistical significance was < 0.05; Mean Difference (Final Values) = -0.002, 95% CI 2-sided [-0.20 to 0.20]

3. Secondary Outcome: Patient Palliative Symptoms Assessment
Description: Patient will be assessed for twelve symptoms (pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being, shortness of breath, constipation, financial distress, and spiritual pain) using a modified Edmonton Symptom Assessment System (ESAS). Each symptom is rated from 0 to 10 on a numerical scale, 0 meaning that the symptom is absent and 10 that it is of the worst possible severity.
Time Frame: Up to 12 weeks after surgery
Population: data were not collected for this outcome measure
Arm/Group | Surgeon-palliative Care Team Co-management (Intervention) | Surgeon Alone Management (Control)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Patient Spiritual Assessment 12 Weeks After Surgery
Description: Patient spiritual symptoms assessment will be assessed using Functional Assessment of Chronic Illness Therapy - Spiritual Well-being (FACIT-Sp-12); 12 item Spiritual Well-being Scale. Score range: 0 to 48; higher scores correspond to better spiritual well-being.
Time Frame: Up to 12 weeks after surgery
Population: Participants with available survey data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Surgeon-palliative Care Team Co-management (Intervention) | Surgeon Alone Management (Control)
Number analyzed (Participants) | 151 | 146
score on a scale | 35.90 (9.40) | 35.89 (8.92)
Statistical Analysis 1: Comparison: Surgeon-palliative Care Team Co-management (Intervention) vs Surgeon Alone Management (Control); Test type: Superiority; p = .997, Regression, Linear — The a priori threshold for statistical significance was < 0.05; Mean Difference (Final Values) = 0.004, 95% CI 2-sided [-2.09 to 2.10] — FACIT-Sp-12 Total Score

5. Secondary Outcome: Patient Prognostic Awareness Assessment Assessment 12 Weeks After Surgery
Description: Patient prognostic awareness is determined based on the Cancer Care Outcomes Research & Surveillance Consortium (CANCORS) study prognostic awareness questions before and after surgery. To each question, the respondent replied Very likely, Somewhat likely, A little likely, Not at all likely, or Don't know.
Time Frame: Up to 12 weeks after surgery
Population: Participants who completed the respective survey questions are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgeon-palliative Care Team Co-management (Intervention) | Surgeon Alone Management (Control)
Number analyzed (Participants) | 137 | 101
Participants
  Help you live longer? (Very likely): number analyzed (Participants) | 101 | 100
  Help you live longer? (Very likely) | 70 | 80
  Help you live longer? (Somewhat likely): number analyzed (Participants) | 101 | 100
  Help you live longer? (Somewhat likely) | 13 | 11
  Help you live longer? (A little likely): number analyzed (Participants) | 101 | 100
  Help you live longer? (A little likely) | 6 | 3
  Help you live longer? (Not at all likely): number analyzed (Participants) | 101 | 100
  Help you live longer? (Not at all likely) | 6 | 3
  Help you live longer? (Don't know): number analyzed (Participants) | 101 | 100
  Help you live longer? (Don't know) | 6 | 3
  Cure your cancer? (Somewhat likely): number analyzed (Participants) | 101 | 101
  Cure your cancer? (Somewhat likely) | 27 | 25
  Cure your cancer? (Very likely): number analyzed (Participants) | 101 | 101
  Cure your cancer? (Very likely) | 39 | 51
  Cure your cancer? (A little likely): number analyzed (Participants) | 101 | 101
  Cure your cancer? (A little likely) | 10 | 10
  Cure your cancer? (Not at all likely): number analyzed (Participants) | 101 | 101
  Cure your cancer? (Not at all likely) | 14 | 10
  Cure your cancer? (Don't know): number analyzed (Participants) | 101 | 101
  Cure your cancer? (Don't know) | 11 | 5
  Help you with problems you were having because of your cancer? (Very likely) | 54 | 57
  Help you with problems you were having because of your cancer? (Somewhat likely) | 54 | 17
  Help you with problems you were having because of your cancer? (A little likely) | 6 | 8
  Help you with problems you were having because of your cancer? (Not at all likely) | 12 | 10
  Help you with problems you were having because of your cancer? (Don't know) | 11 | 9
Statistical Analysis 1: Comparison: Surgeon-palliative Care Team Co-management (Intervention) vs Surgeon Alone Management (Control); Analysis of question "Help you live longer?"; Test type: Superiority; p = .484, Regression, Linear — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: Surgeon-palliative Care Team Co-management (Intervention) vs Surgeon Alone Management (Control); Analysis of question "Cure your cancer?"; Test type: Superiority; p = .343, Regression, Linear — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 3: Comparison: Surgeon-palliative Care Team Co-management (Intervention) vs Surgeon Alone Management (Control); Analysis of question "Help you with problems you were having because of your cancer?"; Test type: Superiority; p = .908, Regression, Linear; The a priori threshold for statistical significance was < 0.05

6. Secondary Outcome: Patient Mortality up to 6 Months
Description: Number of surviving patients in both arms will be reported at end of 6 months.
Time Frame: Up to 6 months after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Surgeon-palliative Care Team Co-management (Intervention) | Surgeon Alone Management (Control)
Number analyzed (Participants) | 171 | 162
Participants
  Alive | 164 | 156
  Died | 7 | 6

7. Secondary Outcome: Caregiver Mood Symptom Assessment at 12 Weeks After Surgery
Description: Caregiver symptoms were measured using the Patient-Reported Outcomes Measurement Information System (PROMIS-29) version 2.1. PROMIS-29 survey questions were each rated on a 5-point Likert scale (range: 1 to 5, higher scores represent a better outcome). Item responses were converted to PROMIS T-scores per the PROMIS scoring manual (population mean = 50, SD = 10). T-scores were then converted to standardized z-scores using the formula (T-score - 50) / 10. Composite physical and mental health z-scores were calculated using weighted domain z-scores. Higher z-scores indicate better outcomes, and negative z-scores indicate scores below the population reference mean.
Time Frame: Up to 12 weeks after surgery
Population: Participants who completed the survey are included in the analysis
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Surgeon-palliative Care Team Co-management (Intervention) | Surgeon Alone Management (Control)
Number analyzed (Participants) | 37 | 40
z-score
  Physical health | 0.32 (0.92) | 0.33 (0.63)
  Mental health | 0.27 (0.94) | 0.23 (0.64)

8. Secondary Outcome: Caregiver Burden Measurement 12 Weeks After Surgery
Description: The Zarit Caregiver Burden Scale (ZBI-12) is a 12-item measure of caregiver burden caring for a patient with chronic illness, focusing on the emotional, physical, and social aspects of caregiving. The questions are ranked on a 5-point Likert scale. The total score is 0-48 a higher score indicates a worse outcome (more caregiver burden).
Time Frame: Up to 12 weeks after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Surgeon-palliative Care Team Co-management (Intervention) | Surgeon Alone Management (Control)
Number analyzed (Participants) | 37 | 40
score on a scale | 6.50 [4.00 to 12.50] | 11.50 [0.75 to 15.75]
Statistical Analysis 1: Comparison: Surgeon-palliative Care Team Co-management (Intervention) vs Surgeon Alone Management (Control); Test type: Superiority; p = .531, Regression, Linear — The a priori threshold for statistical significance was < 0.05

9. Secondary Outcome: Caregiver Spiritual Measure at 12 Weeks
Description: Caregiver spiritual symptoms assessment will be assessed using Functional Assessment of Chronic Illness Therapy - Spiritual Well-being (FACIT-Sp-12); 12 item Spiritual Well-being Scale (score range: 0 to 48; higher scores correspond to better spiritual well-being).
Time Frame: Up to 12 weeks after surgery
Population: Participants with available survey data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Surgeon-palliative Care Team Co-management (Intervention) | Surgeon Alone Management (Control)
Number analyzed (Participants) | 37 | 40
score on a scale | 34.06 (8.34) | 33.72 (7.55)
Statistical Analysis 1: Comparison: Surgeon-palliative Care Team Co-management (Intervention) vs Surgeon Alone Management (Control); Test type: Superiority; p = .871, Regression, Linear — The a priori threshold for statistical significance was < 0.05

10. Secondary Outcome: Caregiver Prognostic Awareness Assessment at 12 Weeks
Description: Caregiver prognostic awareness was determined based on the Cancer Care Outcomes Research & Surveillance Consortium (CANCORS) study prognostic awareness questions before and after surgery. To each question, the respondent replied Very likely, Somewhat likely, A little likely, Not at all likely, or Don't know.
Time Frame: Up to 12 weeks after surgery
Population: Participants who completed the respective survey questions are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgeon-palliative Care Team Co-management (Intervention) | Surgeon Alone Management (Control)
Number analyzed (Participants) | 101 | 100
Participants
  Awareness after: Help your loved one live longer? (Very Likely): number analyzed (Participants) | 101 | 99
  Awareness after: Help your loved one live longer? (Very Likely) | 77 | 83
  Awareness after: Help your loved one live longer? (Somewhat likely): number analyzed (Participants) | 101 | 99
  Awareness after: Help your loved one live longer? (Somewhat likely) | 12 | 7
  Awareness after: Help your loved one live longer? (A little likely): number analyzed (Participants) | 101 | 99
  Awareness after: Help your loved one live longer? (A little likely) | 0 | 3
  Awareness after: Help your loved one live longer? (Not at all likely): number analyzed (Participants) | 101 | 99
  Awareness after: Help your loved one live longer? (Not at all likely) | 8 | 3
  Awareness after: Help your loved one live longer? (Don't know): number analyzed (Participants) | 101 | 99
  Awareness after: Help your loved one live longer? (Don't know) | 4 | 3
  Awareness after: Cure your loved one's cancer? (Very likely) | 39 | 33
  Awareness after: Cure your loved one's cancer? (Somewhat likely) | 23 | 37
  Awareness after: Cure your loved one's cancer? (A little likely) | 8 | 10
  Awareness after: Cure your loved one's cancer? (Not at all likely) | 19 | 10
  Awareness after: Cure your loved one's cancer? (Don't know) | 12 | 10
  Awareness after: Help your loved one with problems due to the cancer? (Very likely) | 58 | 50
  Awareness after: Help your loved one with problems due to the cancer? (Somewhat likely) | 15 | 23
  Awareness after: Help your loved one with problems due to the cancer? (A little likely) | 4 | 7
  Awareness after: Help your loved one with problems due to the cancer? (Not at all likely) | 12 | 10
  Awareness after: Help your loved one with problems due to the cancer? (Don't know) | 12 | 10
Statistical Analysis 1: Comparison: Surgeon-palliative Care Team Co-management (Intervention) vs Surgeon Alone Management (Control); Analysis of question "Help your loved one live longer?"; Test type: Superiority; p = .770, Regression, Linear — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: Surgeon-palliative Care Team Co-management (Intervention) vs Surgeon Alone Management (Control); Analysis of question "Awareness after: Cure your loved one's cancer?"; Test type: Superiority — The a priori threshold for statistical significance was < 0.05; p = .755, Regression, Linear
Statistical Analysis 3: Comparison: Surgeon-palliative Care Team Co-management (Intervention) vs Surgeon Alone Management (Control); Analysis of question "Awareness after: Help your loved one with problems due to the cancer?"; Test type: Superiority; p = .929, Regression, Linear — The a priori threshold for statistical significance was < 0.05

ADVERSE EVENTS:
Time Frame: up to 1 year
Arm/Group | Surgeon-palliative Care Team Co-management | Surgeon Alone Management
All-Cause Mortality (participants affected / at risk) | 7/182 | 6/177
Serious Adverse Events (participants affected / at risk) | 0/182 | 0/177
Other Adverse Events (participants affected / at risk) | 0/182 | 0/177

LIMITATIONS AND CAVEATS:
Over half of the study occurred during the COVID-19 pandemic, with potential pandemic-related impacts. A majority of participants were White and highly educated, and they received care from urban and suburban tertiary or quaternary medical centers; study results may be less generalizable for non-White, less educated, or rural populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/09/NCT03611309/Prot_SAP_000.pdf